CLINICAL TRIAL: NCT02296047
Title: Ventilation-drive Coupling to Evaluate The Efficacy of Inhaled Bronchodilators in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Ventilation-drive Coupling to Evaluate The Efficacy of Inhaled Bronchodilators in Patients With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Collaborators: Guangzhou Panyu Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CX62782296
Record Dates: First submitted 2014-11-10; First posted 2014-11-20 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2014-11

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD, central drive, bronchodilators
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Ipratropium; Albuterol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): The medication order: subjects inhaled placebo,ipratropium bromide 80μg, salbutamol 400μg in sequence.
  Interventions: Drug: Placebo; Drug: ipratropium bromide; Drug: salbutamol
- Group B (Experimental): The medication order: subjects inhaled placebo, salbutamol 400μg, ipratropium 80μg in sequence.
  Interventions: Drug: Placebo; Drug: ipratropium bromide; Drug: salbutamol

INTERVENTIONS:
Drug: Placebo — physiological saline
  Other Names: Physiological Saline 9 mg/ml
Drug: ipratropium bromide — 80 µg inhalation once
  Other Names: atrovent
Drug: salbutamol — 400 µg inhalation once
  Other Names: Ventolin

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a major cause of chronic morbidity, mortality and disability throughout the world, leading to a heavy social and economic burden.Bronchodilators, the most commonly used drugs in COPD patients, have been shown to reduce dyspnea, improve exercise tolerance and improve health status. However,conventional lung function parameters such as forced vital capacity (FVC) and forced expiratory volume in one second (FEV1) frequently fail to detect significant functional responses to bronchodilators in patients with chronic airflow obstruction. It is necessary for clinical and scientific reasons to develop a new tool to objectively assess the effect of different treatments including bronchodilator on COPD. Our previous study showed that Ventilation-drive coupling may be more sensitive and accurate to evaluate the efficacy of inhaled bronchodilators in patients with COPD because it could better reflect the pathological and physiological characteristics of COPD.

Based on the above conclusion, the present study were performed using the experimental methods of placebo and self-controlled. We aimd to explore the value of ventilation-drive coupling in evaluating the efficacy of bronchodilators on COPD and provide a reasonable basis for the clinical application of this index.

DETAILED DESCRIPTION:
Patients were randomly assigned to one of two intervention groups:

1. Group A: Patients inhaled placebo, ipratropium 80μg, salbutamol 400 μg in sequence;
2. Group B: Patients inhaled placebo, salbutamol 400μg, ipratropium 80 μg in sequence.

The data were collected in 30 minutes after patients inhaled placebo,in 30 minutes after ipratropium and in 15 minutes after salbutamol.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 40-70 years old; Patients with pulmonary function test of FEV1/FVC < 70% and FEV1%pred < 50%; Patients in a clinically stable state; Patients who signed informed consent.

Exclusion Criteria:

Patients with signs of an airway infection; Patients with an acute exacerbation during the previous 4 weeks; Patients with giant bulla(≥3cm in diameter); Patients with recent upper abdominal surgery; Patients with one or more of the following diseases: esophageal cancer, reflux esophagitis, severe obstructive sleep apnea (apnea hypopnea index>15/hr), neuromuscular disease, or significant heart failure; Patients with poor compliance.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Diaphragmatic function | The groups will be assessed at baseline (time zero) and ten minutes after using each drug.
  Diaphragmatic function can be assessed by diaphragm electromyogram (EMGdi), which reflect the physiological activity of the diaphragm and indicate functional status of the central drive.

SECONDARY OUTCOMES:
Respiratory pressure | The groups will be assessed at baseline (time zero) and ten minutes after using each drug.
  Respiratory pressure parameters include gastric pressure (Pga), esophageal pressure (Pes), transdiaphragmatic pressure ( Pdi), mouth pressure (Pmo).
Respiratory volume | The groups will be assessed at baseline (time zero) and ten minutes after using each drug.
  Respiratory volume is associated with Flow, Inspiratory capacity (IC), tidal volume (VT), respiratory rate (RR), inspiratory time (Ti),expiratory time (Te), minute ventilation (VE).

OTHER OUTCOMES:
Degree of dyspnea | The groups will be assessed at baseline (time zero) and ten minutes after using each drug.
  Difference in the degree of dyspnea can be measured by Borg index.

CONTACTS AND LOCATIONS:
Overall Officials: Chen Xin, Doctor, Principal Investigator — Zhujiang Hospital,Southern Medical Unversity
Locations (1):
- Zhujiang Hospital,Southern Medical Universtiy, Guangzhou, Guangdong, China